CLINICAL TRIAL: NCT00426166
Title: Assessment of Infrared Photobiotherapy for Improved Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Martin Skie, MD, Principal Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wound Healing
Record Dates: First submitted 2007-01-22; First posted 2007-01-24 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Wound Healing
MeSH Terms: interventions — Low-Level Light Therapy

ARMS (2):
- 1 (Experimental): Low Level Laser Therapy
  Interventions: Device: Low Level Laser Therapy
- 2 (No Intervention): No Laser Therapy. Outcome Measures the same.

INTERVENTIONS:
Device: Low Level Laser Therapy — 7500 megawatts with a 980 nm treatment beam every 48 hours for two weeks beginning at suture removal.
  Arms: 1

SUMMARY:
The purpose of this study is to examine whether or not Low Level Laser Therapy (LLLT) can reduce pain and/or improve wound healing in patients with an acute traumatic injury to the upper extremity (wrist, forearm, or elbow).

DETAILED DESCRIPTION:
This is a prospective, two group, controlled study using random assignment. All eligible patients will be randomly assigned to one of two groups: the control group (usual care) or the experimental group (usual care plus LLLT). We plan to enroll 50 subjects in this study: 25 subjects will be randomly assigned to the LLLT group and 25 to the usual care group.

All subjects will be recruited within one to two days prior to hospital discharge or at the time of their first postoperative clinic visit. No subjects will be recruited while sedated or receiving intravenous pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 85 years
* Acute traumatic injury of an upper extremity (wrist, forearm, or elbow)
* Currently resides within 100 miles of UMC

Exclusion Criteria:

* Pregnant
* Pacemaker
* Medications that have heat or light-sensitivity contraindications (such as: steroids, some antibiotics)
* Two or more cardiac risk factors
* Intraoperative complications
* Wound infection
* Open Wound

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Skie, MD, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per the initial IRB application, the criteria for selection and exclusion was based on the following:
  Inclusion - Adult patients with unhealed wounds of the upper extremity.
  For Outcome Measures, study results were destroyed/shredded based on 3 year minimum record retention after completion of research. Not able to provide patient reported ranges. Only data available is means.
Groups:
- Low Level Laser Therapy Group: Low Level Laser Therapy: 7500 megawatts with a 980 nm treatment beam every 48 hours for two weeks beginning at suture removal.
- Standard Treatment Control Group: No Laser Therapy. Outcome Measures the same.
Period: Overall Study
Arm/Group | Low Level Laser Therapy Group | Standard Treatment Control Group
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Level Laser Therapy Group: Low Level Laser Therapy: Low Level Laser Therapy on Wound
- Total: Total of all reporting groups
Arm/Group | Low Level Laser Therapy Group | Standard Treatment Control Group | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: Participants]
  Unknown gender | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: FACES Pain Rating Scale Scores
Description: The FACES pain scale ranged from 0-10, with lower scores representing less pain and better outcome.
Time Frame: baseline (2 weeks after surgery)
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Low Level Laser Therapy: Low Level Laser Therapy: Low Level Laser Therapy on Wound
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
units on a scale | 2.0 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 3.3 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

2. Primary Outcome: FACES Pain Rating Scale Scores
Description: The FACES pain scale ranged from 0-10, with lower scores representing less pain and better outcome.
Time Frame: 6 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy Group | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 1.0 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 2.5 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

3. Primary Outcome: FACES Pain Rating Scale.
Description: The FACES pain scale ranged from 0-10, with lower scores representing less pain and better outcome.
Time Frame: 12 weeks after surgery
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Low Level Laser Therapy Group | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
units on a scale | 1.0 [NA to NA] — Please note: Study results/data destroyed and not available to report outcome measures due to 3 year minimum record retention. | 1.5 [NA to NA] — Please note: Study results/data destroyed and not available to report outcome measures due to 3 year minimum record retention.

4. Secondary Outcome: 36-Item Short Form Survey - Bodily Pain Scores
Description: Response to questions generates a numerical score, with a higher score representing a better outcome.
  Measures health-related quality of life across 8 domains, with each domain scored on a scale of 0-100 with higher scores representing a better outcome. Items in the same scale are averaged together to create the 8 scale scores.
Time Frame: baseline (2 weeks after surgery)
Measure: Mean (Full Range); unit: Units in a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units in a scale | 45 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 13 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

5. Secondary Outcome: 36-Item Short Form Survey - Bodily Pain Scores
Description: as for outcome 4
Time Frame: 6 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy Group | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 49 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 44 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

6. Secondary Outcome: 36-Item Short Form Survey - Bodily Pain Scale
Description: as for outcome 4
Time Frame: 12 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 45 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 52 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

7. Secondary Outcome: 36-Item Short Form Survey - General Health
Description: as for outcome 4
Time Frame: 2 weeks after surgery (baseline)
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 70 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 54 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

8. Secondary Outcome: 36-Item Short Form Survey - General Health
Description: as for outcome 4
Time Frame: 6 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 75 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 58 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

9. Secondary Outcome: 36-Item Short Form Survey - General Health
Description: as for outcome 4
Time Frame: 12 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 60 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 55 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

10. Secondary Outcome: 36-Item Short Form Survey - Physical Function
Description: as for outcome 4
Time Frame: 2 weeks after surgery (baseline)
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 54 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 52 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

11. Secondary Outcome: 36-Item Short Form Survey - Physical Function
Description: as for outcome 4
Time Frame: 6 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 50 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 70 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

12. Secondary Outcome: 36-Item Short Form Survey - Physical Function
Description: as for outcome 4
Time Frame: 12 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 50 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 63 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

13. Secondary Outcome: 36-Item Short Form Survey - Mental Health
Description: as for outcome 4
Time Frame: 2 weeks after surgery (baseline)
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 59 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 58 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

14. Secondary Outcome: 36-Item Short Form Survey - Mental Health
Description: as for outcome 4
Time Frame: 6 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 58 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 71 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

15. Secondary Outcome: 36-Item Short Form Survey - Mental Health
Description: as for outcome 4
Time Frame: 12 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 60 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 60 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

16. Secondary Outcome: 36-Item Short Form Survey - Social Function
Description: as for outcome 4
Time Frame: 2 weeks after surgery (baseline)
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 55 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 40 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

17. Secondary Outcome: 36-Item Short Form Survey - Social Function
Description: as for outcome 4
Time Frame: 6 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 58 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 84 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

18. Secondary Outcome: 36-Item Short Form Survey - Social Function
Description: as for outcome 4
Time Frame: 12 weeks after surgery
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
Number analyzed (Participants) | 13 | 14
Units on a scale | 58 [NA to NA] — All data related to the study has been destroyed. Only data available is means. | 74 [NA to NA] — All data related to the study has been destroyed. Only data available is means.

ADVERSE EVENTS:
Time Frame: From the time of surgery to 12 weeks post op.
Arm/Group | Low Level Laser Therapy | Standard Treatment Control Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes